CLINICAL TRIAL: NCT03325790
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Safety And Efficacy of SPI-1005 in Meniere's Disease
Brief Title: SPI-1005 for the Treatment of Patients With Meniere's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1005-251
Record Dates: First submitted 2017-10-04; First posted 2017-10-30 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Meniere's Disease
Keywords: Meniere's disease; Hearing Loss; Vertigo; Tinnitus; Ebselen; Pharmacokinetics; Safety; Efficacy; Speech
MeSH Terms: conditions — Meniere Disease; Hearing Loss; Vertigo; Tinnitus; Speech | interventions — ebselen

STUDY DESIGN:
Intervention Model Description: RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: DOUBLE-BLIND
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 200mg SPI-1005 twice daily (BID) (Experimental): 200mg SPI-1005 BID
  Interventions: Drug: 200mg SPI-1005 BID
- 400mg SPI-1005 BID (Experimental): 400mg SPI-1005 BID
  Interventions: Drug: 400mg SPI-1005 BID

INTERVENTIONS:
Drug: 200mg SPI-1005 BID — Active: low dose
  Other Names: ebselen
  Arms: 200mg SPI-1005 twice daily (BID)
Drug: 400mg SPI-1005 BID — Active: high dose
  Other Names: ebselen
  Arms: 400mg SPI-1005 BID
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, efficacy, and Pharmacokinetics (PK) of two dose levels of SPI-1005 administered for 28 days compared to placebo in patients with Meniere's disease.

DETAILED DESCRIPTION:
Study participants will be randomized to SPI-1005 or placebo in this double-blind study to evaluate both safety and efficacy of the investigational treatment. Participants, aged 18-75 years, with probable or definite Meniere's disease will undergo baseline testing to assess severity of sensorineural hearing loss, tinnitus and vertigo. During the study, and 28 days after completion of treatment, participants will be evaluated for safety (adverse events, physical examinations, vital signs and clinical laboratory testing (CBC,serum chemistry). Trough plasma levels of ebselen and its major metabolite will be determined using liquid chromatography-mass spectrometry (LCMS) at specified visits. Additionally, plasma will be analyzed for selenium at the corresponding visits. The effect of SPI-1005 on hearing and balance will be evaluated. Tinnitus (TFI) and vertigo (VSS) will be evaluated at baseline, during and study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, 18-75 years of age at the time of enrollment.
* Diagnosis of probable or definitive Meniere's disease by American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS) 1995 criteria.
* Two of three active symptoms including vertigo or disequilibrium, fluctuating hearing loss, or tinnitus within the 3 months prior to study enrollment.
* Hearing loss of ≥ 30 decibels (dBHL) at either 250, 500 or 1000 Hz.
* Voluntary consent to participate in the study.
* Male subjects that are willing to use condoms throughout the study period and 90-days following study completion even if not fertile.
* Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to screening and throughout the study or be using one of the following acceptable birth control methods:

  * Intrauterine Device in place for at least 3 months prior to study; or
  * Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion; or
  * Stable hormonal contraceptive for at least 3 months prior to study and through study completion; or
  * Surgical sterilization (vasectomy) of partner at least 6 months prior to study enrollment.
* Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study enrollment, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be at least 1 year since last menses.

Exclusion Criteria:

* Current use of or within 60 days prior to study IV ototoxic medications such as chemotherapy including cisplatin, carboplatin, or oxaliplatin; aminoglycoside antibiotics including gentamicin, amikacin, tobramycin, kanamycin, or streptomycin; or loop diuretics including furosemide.
* History of otosclerosis or vestibular schwannoma.
* History of significant middle ear or inner ear surgery.
* Current conductive hearing loss, otitis media, or mixed hearing loss.
* Significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, or psychiatric disease.
* Current use or within 30 days prior to study enrollment systemic steroids or drugs known to be strong inhibitors or inducers of cytochrome P450 enzymes.
* Hypersensitivity or idiosyncratic reaction to compounds related to ebselen or selenium.
* Female patients who are pregnant or breastfeeding.
* Participation in another interventional drug or device study within 30 days prior to study consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kil, MD, Study Chair — Sound Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - Ccent/Cccr, Fresno, California
  - UCSD, San Diego, California
  - UCSF, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - UMiami, Miami, Florida
  - KUMC, Kansas City, Kansas
  - Advanced ENT & Allergy, Louisville, Kentucky
  - ENT and Allergy Associates, LLP, New York, New York
  - CEENTA, Charlotte, North Carolina
  - TJU, Philadelphia, Pennsylvania
  - MUSC, Charleston, South Carolina
  - UT Southwestern, Dallas, Texas
  - Northwest Ear, Inc., Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kil J, Pierce C, Tran H, Gu R, Lynch ED. Ebselen treatment reduces noise induced hearing loss via the mimicry and induction of glutathione peroxidase. Hear Res. 2007 Apr;226(1-2):44-51. doi: 10.1016/j.heares.2006.08.006. Epub 2006 Oct 6. PMID 17030476
- [Background] Lynch E, Kil J. Development of ebselen, a glutathione peroxidase mimic, for the prevention and treatment of noise-induced hearing loss. Semin Hear 2009; 30(1):47-55
- [Background] Kil J, Lobarinas E, Spankovich C, Griffiths SK, Antonelli PJ, Lynch ED, Le Prell CG. Safety and efficacy of ebselen for the prevention of noise-induced hearing loss: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2017 Sep 2;390(10098):969-979. doi: 10.1016/S0140-6736(17)31791-9. Epub 2017 Jul 14. PMID 28716314
- [Background] Kil J, Harruff EE, Longenecker RJ. Development of ebselen for the treatment of sensorineural hearing loss and tinnitus. Hear Res. 2022 Jan;413:108209. doi: 10.1016/j.heares.2021.108209. Epub 2021 Feb 19. PMID 33678494
- [Derived] Nelson L, Johns JD, Gu S, Hoa M. Utilizing Single Cell RNA-Sequencing to Implicate Cell Types and Therapeutic Targets for SSNHL in the Adult Cochlea. Otol Neurotol. 2021 Dec 1;42(10):e1410-e1421. doi: 10.1097/MAO.0000000000003356. PMID 34510123
- See also: Sound Pharmaceuticals, Inc. — http://www.soundpharma.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent screening procedures, including audiometric evaluation, to ensure they met inclusion/exclusion criteria prior to assignment to a treatment group. 20 patients were screen failures due to not meeting specific inclusion/exclusion criteria. 3 patients were eligible for the study and were assigned to an arm/group but did not start treatment.
Period: Overall Study
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Started | 42 | 42 | 42
Completed | 41 | 41 | 38
Not Completed | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID | Total
Number analyzed (Participants) | 42 | 42 | 42 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.03) | 55.9 (9.55) | 50.6 (10.55) | 53.9 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 20 | 66
  Male | 22 | 16 | 22 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 4 | 14
  Not Hispanic or Latino | 39 | 35 | 38 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 39 | 37 | 39 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 42 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: Number and severity of adverse events in patients treated with placebo versus SPI-1005.
  Outcome Measure 1 includes all adverse events, including those which are not reported in the Adverse Event module, i.e., adverse events which did not result in death, were not Serious Adverse Events, and which were below the frequency threshold (5%) in any arm as required for reporting.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 42 | 42 | 42
Participants
  Total Number of Patients with Treatment Emergent Adverse Events (TEAE) | 19 | 20 | 20
  Number of Patients with Mild TEAE | 15 | 18 | 18
  Number of Patients with Moderate TEAE | 6 | 3 | 7
  Number of Patients with Severe TEAE | 0 | 0 | 2

2. Primary Outcome: Efficacy of SPI-1005 on Hearing Loss
Description: Improvement in sensorineural hearing loss from baseline using Pure Tone Audiometry
Time Frame: 8 weeks
Population: Analysis population includes those participants who completed the outcome measure at baseline and 8-week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 41 | 42 | 41
Participants
  Threshold Improvement from Baseline >=10 dB in at least 1 low frequency (250, 500, or 1000 Hz): Yes | 15 | 16 | 25
  Threshold Improvement from Baseline >=10 dB in at least 1 low frequency (250, 500, or 1000 Hz): No | 26 | 26 | 16
  Threshold Improvement >=10 dB in 2 adjacent low frequencies (250 and 500 Hz, or 500 and 1000 Hz): number analyzed (Participants) | 41 | 42 | 40
  Threshold Improvement >=10 dB in 2 adjacent low frequencies (250 and 500 Hz, or 500 and 1000 Hz): Yes | 8 | 7 | 15
  Threshold Improvement >=10 dB in 2 adjacent low frequencies (250 and 500 Hz, or 500 and 1000 Hz): No | 33 | 35 | 25

3. Primary Outcome: Efficacy of SPI-1005 on Word Recognition Score
Description: Improvement in Words-in-Noise (WIN) test score from baseline. WIN test score, 0-35 words, in which a higher score means a better outcome.
Time Frame: 8 weeks
Population: Analysis population includes those participants who completed the outcome measure at baseline and 8-week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 41 | 41 | 40
Participants
  WIN Score Improvement from Baseline >=10%: Yes | 23 | 23 | 30
  WIN Score Improvement from Baseline >=10%: No | 18 | 18 | 10
  WIN Score Improvement from Baseline >=20%: Yes | 19 | 17 | 27
  WIN Score Improvement from Baseline >=20%: No | 22 | 24 | 13
  WIN Score Improvement from Baseline >= 4 words: Yes | 14 | 13 | 24
  WIN Score Improvement from Baseline >= 4 words: No | 27 | 28 | 16

4. Primary Outcome: Efficacy of SPI-1005 on Tinnitus
Description: Improvement in the Tinnitus Functional Index (TFI) from baseline. TFI Total Score: 0-100, in which a higher score means a worse outcome.
Time Frame: 8 weeks
Population: Analysis population includes those participants who completed the outcome measure at baseline and 8-week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 41 | 42 | 41
Participants
  TFI Total Score >= 10pt. reduction from Baseline | 20 | 19 | 13
  No TFI Total Score >= 10pt. reduction from Baseline | 21 | 23 | 28

5. Primary Outcome: Efficacy of SPI-1005 on Tinnitus Loudness
Description: Improvement in Tinnitus Loudness (TL) on response to Tinnitus Functional Index Question Number 2.
  Question Number 2: "How Strong or Loud is your tinnitus?": 0-10, in which a higher score means a worse outcome.
Time Frame: 8 weeks
Population: Analysis population includes those participants who completed the outcome measure at baseline and 8-week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 41 | 42 | 41
Participants
  TL >= 2pt. reduction from Baseline | 14 | 15 | 14
  No TL >= 2pt. reduction from Baseline | 27 | 27 | 27

6. Primary Outcome: Efficacy of SPI-1005 on Vertigo
Description: Improvement in Vertigo Symptom Scale (VSS) from baseline. VSS Total Scale: 0-60, in which a higher score means a worse outcome
Time Frame: 8 weeks
Population: Analysis population includes those participants who completed the outcome measure at baseline and 8-week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 41 | 42 | 41
Participants
  VSS Total Scale >= 6pt. reduction from Baseline | 21 | 21 | 18
  No VSS Total Scale >= 6pt. reduction from Baseline | 20 | 21 | 23

7. Secondary Outcome: Trough Plasma Concentration of SPI-1005
Description: Trough plasma concentration of SPI-1005 (ebselen) will be determined at certain time intervals
Time Frame: 2 weeks, 4 weeks, 8 weeks
Population: In the placebo group, all ebselen concentrations were below the limit of quantitation at all timepoints studied. Therefore, the Analysis Population only includes the SPI-1005 groups.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
Number analyzed (Participants) | 42 | 42
ng/mL
  2 weeks: number analyzed (Participants) | 38 | 37
  2 weeks | 27.2 (19.8) | 48.4 (33.2)
  4 weeks: number analyzed (Participants) | 38 | 37
  4 weeks | 19.7 (14.7) | 40.6 (29.1)
  8 weeks: number analyzed (Participants) | 37 | 38
  8 weeks | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo | 200mg SPI-1005 Twice Daily (BID) | 400mg SPI-1005 BID
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 3/42 | 7/42 | 8/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | 200mg SPI-1005 Twice Daily (BID) (N=42) | 400mg SPI-1005 BID (N=42)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 4 (4)
Blood triglycerides increased (Investigations) | 1 (1) | 5 (5) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will not, during or subsequent to the term of the Clinical Trial Agreement, use Confidential Information for any purpose whatsoever other than the performance of the Services, and will not disclose Confidential Information to any third party. Confidential Information will remain the sole property of Sponsor, as applicable.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT03325790/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03325790/SAP_001.pdf